CLINICAL TRIAL: NCT02771080
Title: Peak Systolic Global Longitudinal Strain and Low Cardiac Output Syndrome After Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Jean François Brichant, Professor, Head of Department, University of Liege
Other Study IDs: CHULgstrain
Record Dates: First submitted 2016-05-11; First posted 2016-05-12 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-06

CONDITIONS: Low Cardiac Output Syndrome After Adult Cardiac Surgery
MeSH Terms: interventions — Cardiac Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Cardiac surgery

SUMMARY:
This is a retrospective observational study to assess the relationship between peak systolic global longitudinal strain measured on pre-cardiopulmonary bypass trans-esophageal echo images predicts post-operative low cardiac output syndrome defined as the need for an inotropic support during 24 hours or longer.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac surgery involving the use of cardiopulmonary bypass
* Availability of pre-cardiopulmonary bypass trans-oesophageal echo images allowing measurement of the peak systolic global longitudinal strain

Exclusion Criteria:

* Preoperative atrial fibrillation
* Preoperative critical state
* Emergent/salvage surgery
* Heart transplant surgery
* Left ventricular assist device implantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing on-pump elective or urgence cardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 275 (Actual)
Dates: Start 2016-06; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Post-operative low cardiac output syndrome | 30 days
  Need for pharmacological inotropic support during 24 hours or more post-operatively

SECONDARY OUTCOMES:
Length of intensive care unit stay | 30 days
Length of hospital stay | 30 days
30-day or in hospital mortality | 30 days
duration of post-operative mechanical ventilation | 30 days
post-operative acute kidney injury | 30 days
Need for readmission to the intensive care | 30 days

REFERENCES:
- [Derived] Amabili P, Benbouchta S, Roediger L, Senard M, Hubert MB, Donneau AF, Brichant JF, Hans GA. Low Cardiac Output Syndrome After Adult Cardiac Surgery: Predictive Value of Peak Systolic Global Longitudinal Strain. Anesth Analg. 2018 May;126(5):1476-1483. doi: 10.1213/ANE.0000000000002605. PMID 29116972